CLINICAL TRIAL: NCT05725447
Title: Cross-cultural Adaptation, Validity and Reliability of the Turkish Version of the Premenstrual Syndrome Impact Questionnaire (PMS-IQ)
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: 83116987-760
Record Dates: First submitted 2023-01-16; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; Turkish version; Translation; Reliability; Validity
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Individuals with premenstrual syndrome
  Interventions: Other: Validity and reliability study

INTERVENTIONS:
Other: Validity and reliability study — Face-to-face questionnaire study

SUMMARY:
This study is aimed to carry out the Turkish version validity and reliability of the Premenstrual Syndrome Impact Questionnaire (PMS-IQ).

DETAILED DESCRIPTION:
Although the severity of premenstrual syndrome (PMS) symptoms varies among women, it is known that PMS symptoms are common, especially in young adult women. The most common symptoms are nervousness, breast tenderness, depression, abdominal swelling and general body edema. Along with personal and mental differences, it has been one of the important problems to cope with PMS symptoms, which are frequently experienced in a variable order from mild to severe in each menstrual cycle period. Sometimes the complaints are so severe that they negatively affect the individual's activities of daily living. This syndrome, which negatively affects the quality of life of the individual, also prepares the ground for the formation of serious mental problems. Most questionnaires for the assessment of premenstrual symptoms only measure the presence and/ or intensity of premenstrual symptoms by a retrospective or prospective grading, not the effect caused by the symptoms. Premenstrual Syndrome Impact Questionnaire (PMS-IQ) assesses functional interaction in daily life as well as psychological stress and is designed for premenstrual symptoms. It takes into account the complex and multifaceted nature of the disorder, thus facilitating the diagnosis process by evaluating the necessary effect and enabling the planning and evaluation of the treatment. There is no Turkish version and validity study of PMS-IQ. This study is aimed to evaluate the validity and reliability of the Turkish version of PMS-IQ. The study of validity and reliability is planned with 99 individuals with PMS. The sociodemographic characteristics of the individuals will be questioned by the investigators and then the patients will be evaluated with PMS-IQ, Premenstrual Coping Measure (PCM), Pain Disability Index (PDI), Big Five Personality Traits Scale (BFPTS), Premenstrual Syndrome Scale (PSS), and Premenstrual Symptoms Impact Survey (PMSIS). The test-retest will be re-administered by face-to-face interview technique after 1 week. The results will be analyzed using the SPSS version 22.0 computer package program.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45
* Meeting the diagnostic criteria for premenstrual dysphoria according to DSM-5
* Not having any diagnosed chronic disease
* Not having past or present mental illness
* Those who can speak, read and write Turkish
* Volunteered to participate in the study

Exclusion Criteria:

* Psychiatric and cognitive impairment such as psychosis, bipolar disorder, eating disorder, moderate or severe depression, or somatic symptom disorder
* Having participated in psychotherapy for premenstrual symptoms (currently or in the past)
* Being pregnant and breastfeeding
* Having acute suicidal tendencies
* Having gynecological diseases (hysterectomy, oophorectomy, gynecological cancer, polycystic ovary syndrome, endometriosis, infertility)
* Using or changing in the past 3 months antidepressants, benzodiazepines/antipsychotics, oral contraceptives or hormones (e.g. thyroid hormones)
* Having any neurological disorder
* Not being able to speak, read or write Turkish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with premenstrual syndrome between the ages of 18-45
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Impact Questionnaire | first and second assessment (baseline and 1 week)
  Premenstrual Syndrome Impact Questionnaire consists of 18 items. It evaluates functional interaction in daily life as well as psychological stress and is designed for premenstrual symptoms. It takes into account the complex and multifaceted nature of the disorder, thus facilitating the diagnosis process by evaluating the necessary effect and enabling the planning and evaluation of the treatment. It has a 4-point Likert-type answer system. The lowest score is 18 and the highest score is 72. The higher the score, the higher the impaction.
Premenstrual Coping Measure | at first assessment (baseline)
  The Premenstrual Coping Measure was developed to assess the ability of Australian women aged 18-49 to cope with premenstrual symptoms. Each item of the five-point Likert-type scale, which consists of 5 sub-dimensions, is scored between 1 and 5. No evaluation is made on the Premenstrual Coping Measure total score. As the score obtained from the sub-dimensions of the scale increases, the ability to cope with premenstrual symptoms also increases. The lowest score is 27, the highest score is 135. Increasing score indicates better coping ability. Turkish version, validity and reliability study of Premenstrual Coping Measure was conducted.
Pain Disability Index | at first assessment (baseline)
  The Pain Disability Index is a self-administered, short and easy scale that measures the extent to which the pain secondary to ongoing discomfort affects the daily life of the individual and the level of disability developed due to this reason. The scale consists of seven questions. The individual is asked to rate the effects of pain on seven functional activities of daily living, consisting of family-home responsibilities, leisure time, occupation, social activity, sexual life, and self-care, by giving a score of 0 to 10 for all questions (0= not prevent, 5=moderate prevents, 10= I'am completely inadequate). The total score ranges from 0 to 70. 40 and above means a high level of disability. High scores indicate that the disability is severe. Turkish version, validity and reliability study is available.
Big Five Personality Traits Scale-10 | at first assessment (baseline)
  Big Five Personality Traits Scale-10 has been brought to the literature as an alternative and short version of Big Five Personality Traits Scale-44. The scale consists of 10 items and 5 sub-dimensions. The scale was evaluated with a 5-point Likert-type rating, as "Strongly Disagree", "Slightly Disagree", "Neither Agree nor Disagree", "Agree Slightly" and "Strongly Agree". The statements numbered 1-3-4-5-7 in the scale were reversed. The lowest score is 10, the highest score is 50. Increasing score and decreasing score according to sub-scales express better and worse personality traits. Turkish version, validity and reliability study of Big Five Personality Traits Scale-10 was conducted.
Premenstrual Syndrome Scale | at first assessment (baseline)
  The Premenstrual Syndrome Scale is a scale that aims to measure the severity of premenstrual symptoms. This scale, which is widely used in Turkey, includes 44 discourses marked by the individual considering "being in the period one week before menstruation". Premenstrual Syndrome Scale with five-point Likert-type consists of 9 sub-dimensions (depressive affect, anxiety, fatigue, irritability, depressive thoughts, pain, appetite changes, sleep changes, bloating). The lowest score that can be obtained from the scale is 44, and the highest score is 220. The sub-dimension scores are obtained by summing the items in these dimensions, and the Premenstrual Syndrome Scale total score is found by the sum of the sub-dimension scores. Those with a Premenstrual Syndrome Scale total score greater than 50% are classified as premenstrual syndrome positive. A higher Premenstrual Syndrome Scale score indicates more severe premenstrual symptoms.
Premenstrual Symptoms Impact Survey | at first assessment (baseline)
  The Premenstrual Symptoms Impact Survey is a 5-point Likert-type scale consisting of 6 items developed as a web-based one to evaluate the impact of premenstrual symptoms on health-related quality of life. As stated in the directive of the scale, to be answered according to the "last premenstrual period"; It has six items on quality of life, including mental health, social functionality, vitality, and role functionality. The evaluation of each substance is made between "1 (no effect)" and "5 (high effect)" according to the degree of impact of the relevant area. The total score of the scale ranges from 6-30, and high scores indicate worsening quality of life. A Turkish validity and reliability study was conducted and it was stated that the scale could evaluate the status and treatment results of PMS in women of reproductive age.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR